CLINICAL TRIAL: NCT06176339
Title: "Assessing the Clinical Utility of Adding Pentoxifylline to Neoadjuvant Chemotherapy Protocols in Breast Cancer Patients"
Brief Title: Assessing the Clinical Utility of Adding Pentoxifylline to Neoadjuvant Chemotherapy Protocols in Breast Cancer Patients"
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Omar Hamdy, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-147-1
Record Dates: First submitted 2023-12-01; First posted 2023-12-19 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Female
Keywords: neoadjuvant chemotherapy; doxorubicin; cyclophosphamide; paclitaxel; efficacy; toxicity
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pentoxyphyllin group (Active Comparator): Patients will undergo a treatment plan determined by the multidisciplinary team. This involves four cycles of intravenous (IV) doxorubicin at a dose of 60 mg/m2 along with IV cyclophosphamide at 600 mg/m2 per cycle. Following this, taxane will be administered. Additionally, patients are prescribed 400 mg pentoxifylline tablets to be taken three times daily.
  Interventions: Drug: Pentoxifylline Oral Tablet
- Control group (Placebo Comparator): Patients will undergo a treatment plan determined by the multidisciplinary team. This involves four cycles of intravenous (IV) doxorubicin at a dose of 60 mg/m2 along with IV cyclophosphamide at 600 mg/m2 per cycle. Following this, taxane will be administered. Additionally, patients will take placebo tablets three times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline Oral Tablet — Pentoxifylline 400 mg extended-release oral tablets will be administered orally three times per day through the chemotherapy cycles.
  Other Names: Intravenous doxorubicin; Intravenous cyclophosphamide; Intravenous taxane
  Arms: Pentoxyphyllin group
Drug: Placebo — Placebo tablets will be administered orally three times per day through the time of the chemotherapy cycles.
  Other Names: Intravenous doxorubicin; Intravenous cyclophosphamide; Intravenous taxane
  Arms: Control group

SUMMARY:
Breast cancer, a leading cause of cancer-related mortality in women worldwide, has spurred the investigation of novel therapeutic approaches. Pentoxifylline (PTX), a synthetic methylxanthine derivative, has shown promise in preclinical studies when combined with conventional anticancer drugs. This study aims to assess PTX's impact when added to neoadjuvant chemotherapy protocols in breast cancer patients, with the goal of improving treatment outcomes and reducing associated toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients >18 years old with histologic confirmation of invasive breast cancer
* Planned to administer neoadjuvant chemotherapy protocol comprised of doxorubicin/ cyclophosphamide followed by paclitaxel (AC/T)
* Adequate hepatic, renal, and bone marrow functions

Exclusion Criteria:

* Patients on treatment regimen of phosphodiesterase inhibitors
* Patients who are taking antiplatelet or anticoagulant treatment
* Patients who are allergic to phosphodiesterase inhibitors
* History of recent hemorrhagic events
* Active peptic ulcer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Relative reduction in tumor size after neoadjuvant chemotherapy treatment | 6 months
  Radiological relative reduction of tumor size (expressed as the largest diameter in millimeters) after completion of neoadjuvant chemotherapy cycles.

SECONDARY OUTCOMES:
The number of patients achieving a pathological complete response | 6 months
  The number of patients achieving a pathological complete response after the completion of neoadjuvant chemotherapy cycles
The relative change of left ventricular ejection fraction (LVEF) | 3 months
  The alterations in left ventricular ejection fraction (LVEF) assessed through echocardiography after four cycles of doxorubicin/cyclophosphamide compared to its baseline level
The incidence of grade 2 or more of neurotoxicity according to common terminology criteria for adverse event (NCI-CTCAE) version 5 | 2 months
  Assessing the grade of neurotoxicity according to common terminology criteria for adverse event (NCI-CTCAE) version 5
The relative change of liver function tests | 6 months
  The change in liver function tests Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), bilirubin level after neoadjuvant chemotherapy compared to their levels at baseline.
The change in Serum Creatinine concentration | 6 months
  The change in Serum Creatinine concentration after neoadjuvant chemotherapy compared to baseline level.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Hamdy Abdelaleem, PhD, Principal Investigator — Oncology Center, Faculty of medicine, Mansoura University
Locations (1):
- Oncology center of Mansoura University, Al Mansurah, Egypt